CLINICAL TRIAL: NCT05739942
Title: Phase Ib Dose Finding Study Assessing Safety and Activity of [177Lu]Lu-NeoB in Combination With Radiotherapy and Temozolomide in Subjects With Newly Diagnosed Glioblastoma and as a Single Agent in Recurrent Glioblastoma
Brief Title: Dose Finding Study of [177Lu]Lu-NeoB in Newly Diagnosed Glioblastoma and in Recurrent Glioblastoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAA603C12101; 2022-502134-10-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-01-17; First posted 2023-02-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Newly Diagnosed and Recurrent Glioblastoma
Keywords: Glioblastoma,; GBM,; Radioligand Therapy,; RLT,; [68Ga]Ga-NeoB,; [177Lu]Lu-NeoB,; Temozolomide,; TMZ,; O-6-methylguanine-DNA methyltransferase,; MGMT
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [177Lu]Lu-NeoB in Combination with Radiotherapy (RT) and Temozolomide (TMZ) (Experimental): In newly diagnosed glioblastoma
  Interventions: Drug: [177Lu]Lu-NeoB; Drug: [68Ga]Ga-NeoB; Other: Temozolomide
- [177Lu]Lu-NeoB as Single Agent (Experimental): In recurrent glioblastoma
  Interventions: Drug: [177Lu]Lu-NeoB; Drug: [68Ga]Ga-NeoB

INTERVENTIONS:
Drug: [177Lu]Lu-NeoB — Radiopharmaceutical solution for infusion
  Other Names: Lu-NeoB
Drug: [68Ga]Ga-NeoB — Either provided as Kit for the radiopharmaceutical preparation of [68Ga]Ga-NeoB or as ready to use radiopharmaceutical solution for injection
  Other Names: Ga-NeoB
Other: Temozolomide — Capsules/ lyophilized powder in single-dose vial for reconstitution.
  Arms: [177Lu]Lu-NeoB in Combination with Radiotherapy (RT) and Temozolomide (TMZ)

SUMMARY:
This study will investigate different doses of [177Lu]Lu-NeoB in combination with RT and TMZ in participants with newly diagnosed glioblastoma, with methylated or unmethylated promoter, to assess the safety and efficacy of [177Lu]Lu-NeoB in combination with the SoC and in recurrent glioblastoma as single agent, to identify the recommended dose and to also explore the safety of the PET imaging agent [68Ga]Ga-NeoB and characterize its uptake in the tumor area.

DETAILED DESCRIPTION:
Newly diagnosed glioblastoma:

Glioblastoma is the most common and aggressive type of primary brain tumor, with a high mortality rate. The current standard of care (SoC) in newly diagnosed glioblastoma includes the combination of the alkylating agent Temozolomide (TMZ) with Radiotherapy (RT). The hypothesis of this study is to improve the outcome for participants by combining the current standard of care with the radioligand therapy [177Lu]Lu-NeoB. Participants with newly diagnosed glioblastoma enrolled into this trial will be treated with the standard regimen TMZ and RT, combined with [177Lu]Lu-NeoB every 4 weeks (Q4W) for 6 administrations. In cases where participants tolerate and benefit from [177Lu]Lu-NeoB, they can receive an additional 4 doses (total up to 10 dose administrations). During this period, regular safety and efficacy assessments are planned on a weekly basis. The primary objective of this trial is to identify the recommended dose of [177Lu]Lu-NeoB in combination with TMZ and RT in participants with newly diagnosed glioblastoma and to characterize the safety and tolerability of this treatment. For this reason, participants will be enrolled and treated in cohorts with increasing dose levels and the totality of available data will be used to define the recommended dose. Contrast enhanced MRI assessments are to be repeated every 8 weeks. Following treatment, all participants will be followed for up to 5 additional years for safety, progression of disease and survival. Participants with newly diagnosed glioblastoma will undergo a baseline [68Ga]Ga-NeoB PET/CT or PET/MRI after the surgery/biopsy of the tumor.

Recurrent glioblastoma:

Participants with recurrent glioblastoma carry a dismal prognosis and a short survival. The primary objective in recurrent glioblastoma is to determine the recommended dose of [177Lu]Lu-NeoB as single agent and to characterize the safety and tolerability of this treatment. For this reason, participants will be enrolled and treated in cohorts with increasing dose levels and the totality of available data will be used to define the recommended dose. In this study, all participants with recurrent glioblastoma will undergo [68Ga]Ga-NeoB PET scan to assess GRPR expression during the screening period. [177Lu]Lu-NeoB will be administered as a single dose every 3 weeks (Q3W) for 6 administrations. Up to 4 additional administrations of [177Lu]Lu-NeoB may be considered if participants tolerate and benefit from [177Lu]Lu-NeoB (total up to 10 dose administrations).

ELIGIBILITY:
Key Inclusion Criteria/Common Criteria (Group 1 - Newly diagnosed glioblastoma, Group 2 - Recurrent glioblastoma):

1. Signed informed consent must be obtained prior to participation in the study
2. Age >= 18 years
3. Histologically confirmed glioblastoma according to WHO classification established following either a surgical resection or biopsy
4. Participants who are receiving corticosteroid treatment with dexamethasone, must be treated with a dose of =<4 mg/day (or other corticosteroids at equivalent dose) for a minimum of 7 days before initiation of study treatment
5. Adequate bone marrow and organ function as defined by the following laboratory values obtained prior to receiving the first study treatment:

   1. Absolute Neutrophil Count (ANC) >= 1.5 x 10^9/L
   2. Platelet count >= 100 x 10^9/L
   3. Hemoglobin >= 10.0 g/dL
   4. Creatinine clearance >= 60 mL/min calculated by the CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) creatinine equation .
   5. Aspartate transaminase (AST) or Alanine transaminase (ALT) =< 3.0 x ULN
   6. Total bilirubin (TBIL) < 1.5 × ULN (any elevated bilirubin should be asymptomatic at enrollment) except for participants with Gilbert's syndrome who may only be included if the total bilirubin is =< 3.0 × ULN or direct bilirubin =< 1.5 × ULN
   7. Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - =< 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis

Key Inclusion Criteria/Newly diagnosed glioblastoma (Group 1):

9. Availability of tumor tissue representative of glioblastoma from definitive surgery or biopsy, to support biomarker analysis 10. Presence of gadolinium enhancement at the tumor region in the pre-surgery MRI

Key Inclusion Criteria/Recurrent glioblastoma (Group 2) 11. Presence of [68Ga]Ga-NeoB uptake by PET/CT or PET/MRI at the tumor region 12. Having first or second glioblastoma recurrence, after standard therapy that includes prior radiation therapy (RT) and at least 12 weeks from completion of RT 13. Evidence of recurrent disease (RD) demonstrated by disease progression using modified Response Assessment in Neuro-Oncology (mRANO) criteria. RD must be documented with at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, according to mRANO criteria. For those participants who will undergo a second surgery for recurrence, pre-surgery MRI will be used for confirmation of RD.

14. If a second surgery is performed for glioblastoma recurrence, the following criteria must be met:

1. residual and measurable disease post-surgery is not required but surgery must have confirmed the recurrence diagnosis by MRI.
2. surgery completed at least 2 weeks prior to study treatment initiation, with post-surgery recovery without any complications related to surgical procedure.

Key Exclusion Criteria/Common Criteria (Group 1 - Newly diagnosed glioblastoma, Group 2 - Recurrent glioblastoma):

1. Additional, concurrent, or active therapy for glioblastoma outside of the present study 4. History or current diagnosis of impaired cardiac function, clinically significant cardiac disease, or ECG abnormalities indicating significant risk of safety for study participants such as:

a. Documented myocardial infarction (MI), angina pectoris, cardiomyopathy, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to study entry b. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following: i. Risk factors for Torsade de Pointes (TdP) including uncorrected hypocalcemia, hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia ii. Concomitant medication(s) with a known risk to prolong the QT interval and/or known to cause Torsade de Pointes that cannot be discontinued or replaced by safe alternative medication (e.g., within 5 half-lives or 7 days prior to starting study drug) iii. Inability to determine the Fridericia QT correction formula (QTcF) interval c. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third-degree AV block) d. Resting QTcF >= 450 msec (male) or >= 460 msec (female) e. Left Ventricular Ejection Fraction (LVEF) <50% as determined by echocardiogram (ECHO) or Multiple Gated Acquisition (MUGA) scan f. Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) >=160 mmHg and/or Diastolic Blood Pressure (DBP) >=100 mm Hg, with or without anti-hypertensive medication.

5. History of another active malignancy in the previous 3 years prior to study entry, except participants with prior history of superficial bladder cancer, any in situ carcinoma or basal or squamous cell skin cancer treated curatively

Key Exclusion Criteria/Newly diagnosed glioblastoma (Group 1):

17. Any prior treatment for glioma of any grade, including: prolifeprospan 20 with carmustine wafer, intracerebral agent, radiation treatment, chemotherapy or immunotherapy

Key Exclusion Criteria/Recurrent glioblastoma (Group 2) 18. Previous treatment with bevacizumab for the treatment of glioblastoma with therapeutic intent, or with bevacizumab as supportive therapy (e.g., edema reduction) within 60 days of initiation of study treatment 19. More than two prior lines of systemic therapy, more than one surgical resection for recurrent disease and treatment with an intracerebral/intracranial agent prior to starting [177Lu]Lu-NeoB. Administration in adjuvant setting counts as a line of prior systemic treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of Dose Limiting Toxicity (DLTs) | Up to 8 weeks (newly diagnosed glioblastoma (GBM)) or 6 weeks (recurrent GBM) after the first administration of [177Lu]Lu-NeoB
  A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness/injury, or concomitant medications that occurs within the DLT observation period of [177Lu]Lu-NeoB. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 5.0 will be used for all grading.
  In Group 1 (newly diagnosed GBM), the DLT observation period is defined as a total of 8 weeks (56 days) from the first administration of [177Lu]Lu-NeoB, to cover the entire duration of concomitant RT and TMZ combination with the first two administrations of [177Lu]Lu-NeoB.
  In Group 2 (recurrent GBM), the DLT observation period is 6 weeks (42 days) starting from the first administration of [177Lu]Lu-NeoB (at Week 1 Day 1) and accounting for assessment of the safety profile during 2 full cycles of [177Lu]Lu-NeoB.

SECONDARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) and serious Adverse Events (SAEs), changes in laboratory parameters, vital signs and Electrocardiogram (ECGs) | From date of enrollment till 28 days after end of Treatment, assessed up to approximately 17 months
  The distribution of adverse events will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Absorbed radiation doses of [177Lu]Lu-NeoB in organs and tumor lesions | Cycles 1, 3 and 5: Day 1 (1-4 hours post-dose/post-infusion (p.i.)), Day 2 (24 hours p.i), Day 3 (48 hours p.i), Day 8 (168 hours p.i) (1 cycle = 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  The [177Lu]Lu-NeoB absorbed dose by body organs and tumor lesions will be determined by calculation of TACs obtained from the radiotracer uptake (as percentage of injected dose) in selected organs and lesions (coming from image quantification).
Concentration of [177Lu]Lu-NeoB in blood over time | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Blood concentration of [177Lu]Lu-NeoB will be summarized with descriptive statistics.
Observed maximum blood concentration (Cmax) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Cmax will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Tmax will be listed and summarized using descriptive statistics.
Area under the blood concentration-time curve (AUC) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. AUC will be listed and summarized using descriptive statistics.
Total systemic clearance for intravenous administration (CL) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. CL will be listed and summarized using descriptive statistics.
Volume of distribution during the terminal phase following intravenous elimination (Vz) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. Vz will be listed and summarized using descriptive statistics.
Terminal half-life (T^1/2) of [177Lu]Lu-NeoB | Cycle 1: Day1 (Pre-dose (before start of infusion), end of infusion, 0.5, 1, 2, 4 and 6 hours (hr) post-dose/post-infusion (p.i.)), Day2 (24 hr p.i), Day3 (48 hr p.i), Day8 (168 h p.i) (1 cycle= 3 weeks (recurrent GBM) or 4 weeks (newly diagnosed GBM))
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization of [177Lu]Lu-NeoB. T^1/2 will be listed and summarized using descriptive statistics.
Progression-free survival (PFS) | From date of first dose to date of confirmed progression, assessed up to approximately 17 months
  PFS is defined as the time from the date of first dose to the date of confirmed progression according to modified RANO or death due to any cause. If no PFS event is observed, PFS will be censored at the date of the last adequate tumor assessment prior to data cut-off date and start of new anti-neoplastic therapy, whichever comes first.
Overall Survival (OS) | From date of first dose to date of death due to any cause, assessed up to approximately 17 months
  OS is defined as the time from date of first dose to date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date).
Incidence and severity of AEs following [68Ga]Ga-NeoB administration | At date of screening and every 8 weeks until disease progression.
  Incidence and severity of AEs following [68Ga]Ga-NeoB administration at screening will be done via the analysis of frequencies for Adverse Event (AEs), Serious Adverse Event (SAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (7):
  - University of California LA, Los Angeles, California
  - University of Colorado Denver, Aurora, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - Univ Hosp Cleveland Medical Center, Cleveland, Ohio
  - Uni of Utah Huntsman Cancer Inst, Salt Lake City, Utah
- France (2):
  - Novartis Investigative Site, Dijon, Cote D Or
  - Novartis Investigative Site, Marseille
- Germany (4):
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rostock
- Novartis Investigative Site, Jerusalem, Israel
- Novartis Investigative Site, Reggio Emilia, RE, Italy
- Novartis Investigative Site, Porto, Portugal
- Spain (5):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No